CLINICAL TRIAL: NCT04928989
Title: What Does Web-based Neck-specific Exercise Add to a Digital Convergence Dialogue Meeting Promoting the Work Situation for Employees With Neck Pain?
Brief Title: Convergence Dialogue Meeting With or Without Neck-specific Exercise Promoting Work Ability
Acronym: WORKCIT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anneli Peolsson, Professor, PhD, MSc PT, MSc HRMD, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-00373
Record Dates: First submitted 2021-06-02; First posted 2021-06-18 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-04

CONDITIONS: Workplace
Keywords: Neck pain; Workplace; Counceling; Exercise; Internet-based intervention
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization will take place from a computer-based generated randomization list developed by a statistician. Randomization will be handled by a person not involved in intervention or evaluation. Investigators/ asessors will be blinded for randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convergence dialogue meeting (Active Comparator): Digital counceling with convergence dialogue tripartite meeting. will be conducted in accordance with work dialogue for return to work. Workplace dialogue among employee with neck problems, an expert in the work environment, and the immediate manager. The purpose of the conversations is, in open dialogue, to reach a common understanding of the situation and identify possible interventions to maintain or improve the employee´s work ability.
  Interventions: Other: convergence dialogue meeting
- Neck-specific exercise in addition to convergence dialogue meeting (Experimental): Neck-specific exercise with digital web-based support and four visits to a physiotherapist. Neck-specific exercise will be performed based on a well-structured framework of neck-specific exercise for facilitation of deep neck muscles, increased muscle coordination, improved neck posture and increased neck muscle endurance. Plus additional convergence dialogue meeting as treatment arm no 1.
  Interventions: Other: convergence dialogue meeting

INTERVENTIONS:
Other: convergence dialogue meeting — Digital counceling with convergence dialogue tripartite meeting. will be conducted in accordance with work dialogue for return to work. Workplace dialogue among employee with neck problems, an expert in the work environment, and the immediate manager. The purpose of the conversations is, in open dialogue, to reach a common understanding of the situation and identify possible interventions to maintain or improve the employee´s work ability.

SUMMARY:
The study will be conducted at workplaces, where the work environment and tasks increase employee risk of developing neck problems. A total of 320 participants will be recruited consecutively and after informed consent randomized to convergenge dialogue meeting with or without neck-specific exercise. The main outcome measure is work ability, measured via the Work Ability Score.

DETAILED DESCRIPTION:
Background: Collaboration between employees, manager and occupational health expert is needed to promote work ability. One effective method is a convergence dialogue meeting (CDM). Based on the existing work situation, factors are identified in these meetings that can strengthen the employee's work ability and opportunities for a sustainable working life. A combination of workplace and individual interventions is recommended for best effect. Neck-specific exercise (NSE) is the method with the most evidence for neck problems. NSE in evidence based form has not been investigated for work-related neck pain. More knowledge is needed regarding how CDM can be combined with NSE because clear guidelines are lacking on the best intervention for increased work ability in the case of neck problems. Also lacking are evaluations of digitally distributed CDMs and NSE with support from a web-based program for the current population. The aim of the proposed randomized controlled study is to investigate the contribution of NSE with four visits to a physiotherapist and support from a web-program in addition to three digital CDMs promoting the work situation.

Methods: The study will be conducted at workplaces, where the work environment and tasks increase employee risk of developing neck problems. A total of 320 participants will be recruited consecutively and after informed consent randomized to CDM with or without NSE. The main outcome measure is work ability, measured via the Work Ability Score. Secondary outcome measures are pain, function, health-related quality of life, work absenteeism and presenteeism, work-related factors, and cost-effectiveness. Pathophysiological aspects regarding inflammation and stress markers measured in blood and saliva will be studied, as will muscular changes measured by microdialysis. Interviews are planned with both employees and managers.

Discussion: The goal of the study is to contribute to improved rehabilitation, strengthened work ability, and a sustainable working life for employees with neck problems.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported neck problems that the person experiences as troublesome, affecting ability to perform work, and lasting at least 4 weeks.
* Neck problems as being predominant.
* Current neck pain ≥ 3 on the numeric rating scale (0-10) [53, 55].
* Persons of working age, 18-65 years, who have a permanent job.
* Neck problems clinically verified through a clinical examination to ensure study criteria are met.
* Answers the baseline questionnaire and attends the first intervention visit.
* Confirms being motivated to participate and completes and signs informed consent, including approval, to contact their immediate supervisor regarding a CDM.

Exclusion Criteria:

* Red flags and illness/injury that are contraindicated for or hinder exercise or may be confounding factors for the results, such as severe cardiovascular/lung disease, malignancy, severe rheumatic disease, severe neurological disease, spinal cord injury, diagnosed severe mental illness, drug or alcohol abuse, neck surgery, neck fracture or dislocation, severe cervical radiculopathy, myelopathy, general body pain (e.g., fibromyalgia, Ehlers-Danlos syndrome, generalized osteoarthritis).
* Known pregnancy.
* Cannot understand/communicate in Swedish and thus would be unable to understand information in the study.

For blood samples (not wanting to participate does not constitute exclusion for the randomized controlled trial), the following exclusion criteria are added: increased tendency to bleed and use of blood thinners.

For the subgroup for microdialysis (n = 30, consecutively asked, 15 persons/group; not wanting to participate does not constitute exclusion for the randomized controlled trial), the following exclusion criteria are added:

* Patients who cannot imagine refraining from non-steroid anti-inflammatory drugsduring 2 days before microdialysis may not participate in the microdialysis part of the study.
* Hypersensitivity to anesthetic and antibiotics.
* Increased tendency to bleed and use of blood-thinning drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Work Ability Score | Change in work Ability Score from baseline, to every month until the 15 month follow-up
  Current work ability compared to when it was at its best

SECONDARY OUTCOMES:
Intensity of pain and bothersomeness | change from baseline to 3 month and 15 month follow-up
  neck pain intensity and bothersomeness, headache intensity on a numeric ratin scale.
Frequency of pain, symtoms and medications | change from baseline to 3 month and 15 month follow-up
  Frequency of pain, pain medication, neck stiffness, numbness/tingling into the arms, having problems lifting the arms, dizziness, sleep, concentration
Neck specific function | change from baseline to 3 month and 15 month follow-up
  Neck Disability Index
Symptom satisfaction | change from baseline to 3 month and 15 month follow-up
  Symptom satisfaction according to Cherkin
Exercise/physical activity level | change from baseline to 3 month and 15 month follow-up
  Exercise/physical activity level
Health related quality of life | change from baseline to 3 month and 15 month follow-up
  EQ-5D-3L
Fear avoidance | change from baseline to 3 month and 15 month follow-up
  Fear avoidance beliefs questionnaire
self rated function | change from baseline to 3 month follow-up
  Patient Specific Functional Scale
work situation | description and change from baseline to 3 month and 15 month follow-up
  description of work tasks
self-rated work situation regarding working hours | description and change from baseline to 3 month and 15 month follow-up
  working hours
perceived exertion at work | change from baseline to 3 month and 15 month follow-up
  Borg ratings of perceived exertion
Work ability | change from baseline to 3 month and 15 month follow-up
  work ability index
Sick leave, | change from baseline to 3 month and 15 month follow-up
  sick leave numbers of days/ month
Presenteeism | change from baseline to 3 month and 15 month follow-up
  presenteeism number of days/ month and Stanford presenteeism scale
Effort-Reward Imbalance | change from baseline to 3 month and 15 month follow-up
  Effort Reward Imbalance questionnaire
Demand-control, support | change from baseline to 3 month and 15 month follow-up
  Swedish Demand Control Support Questionnaire which is a short version of the Job centent questionnaire
Risk identifaction at work | change from baseline to 3 month and 15 month follow-up
  Structured multidisciplinary work evaluation tool
work adaptation | change from baseline to 3 month and 15 month follow-up
  work adaptation such as self strategies to be able to work
Time sitting | change from baseline to 3 month and 15 month
  Time sitting at work and during leisure time
Anxiety and depression | change from baseline to 3 month and 15 month follow-up
  Hospital Anxiety and Depression scale
Overall outcome | change from baseline to follw-ups at 3 month and 15 month
  Global rating of change scale
Fulfilment of treatment expectation | 3 month and 15 month related to the patient own expectations
  Fulfilment of treatment expectation, have your expectations been fulfilled: yes, yes partly, no
Satisfaction with the caregiver visits in the study | 3 month, 15 month
  Patient enablement questionnaire
Adverse events/ side-effects | 3 month, 15 month
  adverese events/ side effects of treatment in the study
Cost-effectiveness | From the time period between baseline to 15 month follow-up
  Cost effectiveness through calculation of direct costs; quantity and type of care (inside and outside the study also including drugs related to pain) from registers and from questionnaires, indirect costs;mainly production loss from registers and from questionnaire.
Saliva samples and blood samples | change from baseline to 3 month in a subgroup of the RCT population, all those who agree and are without contra indication
  Inflammation markers, stress markers. The samples will be taken in the morning on an empty stomach. Saliva will be collected with Salivette. Venous blood samples (10-20 ml) from the elbow fold will be collected in EDTA tubes. identification and quantification of proteins.
Microdialysis, tissue changes in the middle Trapezius | baseline, 3 month, subgroup of the RCT population approximately n=30
  Biomechanical changes interstitialli in M. Trapezius. Through microdialysis technology, it is possible to monitor biochemical changes interstitially in the tissue. The technique involves the exchange of substances via diffusion between the tissue and a diaphragmatic catheter inserted into the tissue and flushed by a fluid (perfusate) that is similar in chemical composition to the fluid in the muscle interstitium.
Interview study of employers | 3 month, subgroup of the RCT population, n=20 approximately
  employers experience with interventions and their impact on work ability, health and work situation
Interview with managers | 3 month, approximately n=20
  Interviews with managers regarding the experience of the convergence dialogue meeting
Observation study | During the 3 month treatment period at tripartiate convergence dialogue meeting
  Observation study regarding the interaction between the participants in the converge dialogue meeting. Qualitative data in natural clinical settings of CDMs will be collected through video recordings (≈ 20) to find the meaning of what happen and the interactions during the dialogue. Tripartiate dialogue between patient, manager and care giver regarding the work situation and how to improve it.
Health related quality of life on vertical visual analogue scale | change from baseline to 3 month and 15 month follow-up
  EQ thermometer
self-rated work situation regarding stress at work | description and change from baseline to 3 month and 15 month follow-up
  work stress
self-rated work situation regarding work environment | description and change from baseline to 3 month and 15 month follow-up
  work environment
self-rated work situation regarding satisfaction at work | description and change from baseline to 3 month and 15 month follow-up
  workplace and work satisfaction
self-rated work situation regarding self-rated work performance | description and change from baseline to 3 month and 15 month follow-up
  work performance
self-rated work situation regarding neck position at work | description and change from baseline to 3 month and 15 month follow-up
  neck position

OTHER OUTCOMES:
profession | baseline
  Swedish standard for work classification
Background data | baseline
  Age, gender, education, family situation, pain duration, expectations, smoking history
ICD 10 code | baseline
  ICD 10 code decided after a physical examination
Pain screening | baseline
  Örebro musculoskeletal pain screeing questionnaire
screening for "yellow flags"- behaviour factors at risk | baseline
  START neck screening tool
Treatment outside the study | 3 month, 15 month
  treatment outside the study
profession, open question | description and change from baseline, 3 month and 15 month follow-up
  open question regarding profession

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Anneli Peolsson, Linköping, Östergötland County
  - Dep. Medical and Health Sciences, Physiotherapy, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No
The data is protected by the Swedish health secrets acts and the European General Data Protection Regulation. Data will be presented on a group level without possibility for individual identification.